CLINICAL TRIAL: NCT03958136
Title: Prediction in Silico of Overall Survival in a Pilot Prospective Cohort Study of Metastatic Breast Cancer Patients
Brief Title: Clinico-biological Data Collection Study of Metastatic Breast Cancer
Acronym: EPICURE_SEIN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: European Regional Development Fund (Other); AstraZeneca (Industry); Novartis (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ICO-N-2017-12
Record Dates: First submitted 2018-12-31; First posted 2019-05-21 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; first metastatic setting; prospective clinico-biological database; multi omic analysis; prediction in silico; overall survival; progression free survival; predictive factors; treatment response; resistance to cancer therapy; socio demographic profile
MeSH Terms: conditions — Breast Neoplasms | interventions — Urination; Patient Reported Outcome Measures

STUDY DESIGN:
Intervention Model Description: monocentric, open, prospective database with specific biopsy and blod collections done (biocollection)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Patients HR + and HER2- (Experimental): At each disease progression, patient will have specific interventions :
  * Metastasis biopsy
  * Biomarkers blood, urine and microbiota samples
  * Patient Reported Outcome (PRO)
  Interventions: Procedure: Metastasis biopsy; Biological: Biomarkers blood, urine and microbiota samples; Behavioral: Patient Reported Outcome (PRO)
- Patients HER2 + with or without HR+ (Experimental): At each disease progression, patient will have specific interventions :
  * Metastasis biopsy
  * Biomarkers blood, urine and microbiota samples
  * Patient Reported Outcome (PRO)
  Interventions: Procedure: Metastasis biopsy; Biological: Biomarkers blood, urine and microbiota samples; Behavioral: Patient Reported Outcome (PRO)
- Patients triple negative (HR- and HER2-) (Experimental): At each disease progression, patient will have specific interventions :
  * Metastasis biopsy
  * Biomarkers blood, urine and microbiota samples
  * Patient Reported Outcome (PRO)
  Interventions: Procedure: Metastasis biopsy; Biological: Biomarkers blood, urine and microbiota samples; Behavioral: Patient Reported Outcome (PRO)

INTERVENTIONS:
Procedure: Metastasis biopsy — Metastasis biopsy will be performed for multi-omic analysis
Biological: Biomarkers blood, urine and microbiota samples — Biomarkers blood, urine and microbiota samples for multi-omic analysis
Behavioral: Patient Reported Outcome (PRO) — Patient Reported Outcome (PRO) will be collected throughout the study duration to assess quality of life, anxiety, depression distress, physical activity and food habits.

SUMMARY:
RATIONALE : Currently, the mechanisms associated with the response or resistance to treatment are poorly understood and are multifactorial. These mechanisms involve clinical and biological factors associated with the host and the tumor and possibly the patient's psycho-social environment.

PURPOSE : This trial will assess the use of a prospective database dedicated to patients with breast cancers that contains clinical data as well as epidemiological, psychological, emotional, social, imaging, biological and bio-pathological data. These data will allow a creation of new modelling algorithms in order to predict response and resistance to treatment.

DETAILED DESCRIPTION:
This prospective study will be conducted on first line metastatic breast cancer patients.

Three phenotypic groups are identified on immunohistochemistry done at inclusion: on metastatic sites or breast tumor if local recurrence, usual treatment protocols are often guided by the following groups:

* Group 1 : Patients HR (Hormon Receptor) + (E (Estrogen Receptor) + and/or PR (Progesterone Receptor) +) and HER2- (Human Epidermal Growth Factor Receptor-2)
* Group 2 : Patients HER2 + with or without HR+
* Group 3 : Patients triple negative (HR- and HER2-) Patients will receive treatments as per standard care according to the patient group.

Standard treatments recommended for treatment first line are:

1. For group 1 : For HR + and HER2- patients :

   * For patients requiring Chemotherapy (visceral crisis), the recommended treatment is : Taxanes based chemotherapy Anthracyclines based chemotherapy
   * For the patients without visceral crisis: the recommended treatment is : Hormonal therapy combined with CDK 4-6 inhibitors (Cyclin-dependent kinase) as recommended in standard care.
2. For group 2 : HER2 + (with or without HR+), the recommended treatment is :

   * Paclitaxel (Taxol) combined with Trastuzumab (Herceptin) and Pertuzumab (Perjeta) as per the institutional standard of care.
   * Docetaxel (Taxotere) combined with Trastuzumab (Herceptin) and Pertuzumab (Perjeta) as per the institutional standard of care.
3. For group 3 : triple negative (HR- and HER2-) patients, the recommended treatment is :

   * Paclitaxel (Taxol) with or without Bevacizumab (Avastin) as per the institutional standard of care.

Further treatment lines are administered according to standard practice. Biological and histological assessments are performed on specific metastasis biopsy samples done at baseline and at each progression.

Physical exam, standard laboratory tests, imaging (CT (computerized tomography) scan, PET-CT (Positron emission tomography-computed tomography) and bone scan (for patients with bone metastasis) will be performed every 2 to 6 months according to patient group.

Clinical, biological, pathological, epidemiological, socio-economic and multi-omic data will be collected throughout the study duration.

These massive data will be used to create new algorithms in order to help clinicians to predict treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the patient prior to performing any protocol-related procedures, including screening biopsy, blood sample, faeces and questionnaires
2. Women > 18 years old at time of written consent
3. Patient with histologically confirmed breast cancer
4. Breast cancer metastatic disease or locally advanced not eligible for local curative treatment intent with or without personal history of adjuvant therapy for this cancer (chemotherapy, radiotherapy, surgery …)
5. Patient with metastases that can be biopsied.
6. Performance status ≤ 2 (according to WHO criteria)
7. Indication of any systemic therapeutic strategy can be performed alongside this current cohort in accordance with national and / or international recommendations.
8. HR and HER2 status on metastatic sites or breast tumor if local recurrence:

   * For group 1 :

     * Histologic and/or cytological confirmation of estrogen-receptor positive (ER+) and/ or progesterone receptor positive (PR+) breast cancer determined by local laboratory testing
     * No HER2-overexpression in the patient's tumor tissue determined by local laboratory testing
   * For group 2 :

     * Histologic and/or cytological confirmation of estrogen-receptor positive or negative and/ or progesterone receptor positive or negative breast cancer determined by local laboratory testing
     * HER2-overexpression in the patient's tumor tissue determined by local laboratory testing
   * For group 3 :

     * Histologic and/or cytological confirmation of estrogen-receptor negative and progesterone receptor negative breast cancer determined by local laboratory testing
     * No HER2-overexpression in the patient's tumor tissue determined by local laboratory testing
9. Menopausal status : as per the institutional standard of care
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
11. Patient must be affiliated to a Social Health Insurance

Exclusion Criteria:

1. Other malignancy treated within the last 5 years (except non-melanoma skin cancer or in situ carcinoma of the cervix)
2. Coagulopathy or other pathology that contraindicates biopsy procedures
3. Prior systemic treatment in metastatic setting
4. Patients with exclusive brain metastasis not available for surgery
5. Pregnant or nursing patient
6. Individual deprived of liberty or placed under the authority of a tutor
7. Impossibility to submit to the medical follow-up of this clinical trial for geographical, social or psychological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Estimated)
Dates: Start 2018-12-24 (Actual); Primary Completion 2035-12-24 (Estimated); Study Completion 2036-12-30 (Estimated)

PRIMARY OUTCOMES:
Creation of complex prospective clinico-biological database in metastatic breast cancer | At each progressive disease, 15 years after inclusion
  specific metastatic biopsy intervention
Creation of complex prospective clinico-biological database in metastatic breast cancer | At each progressive disease, 15 years after inclusion
  search of algorithms combining multiple data (clinical, biological, imaging) in breast cancer management
Overall survival | 15 years after inclusion
  Overall Survival is the delay between the date of inclusion and the date of death or last follow-up assessment if censored.

SECONDARY OUTCOMES:
Progression free survival | 15 years after inclusion
  Progression Free survival is the delay between the first dose of a treatment sequence and the date of documented disease progression or death
Quality of life during treatment | every 4-6 months for 15 years after inclusion
  QLQ-C30 Questionnaire (total score)
Quality of life during treatment | every 4-6 months for 15 years after inclusion
  BR23 Questionnaire (total score)
Quality of life during treatment | every 4-6 months for 15 years after inclusion
  STAI anxiety Questionnaire (total score)
Quality of life during treatment | every 4-6 months for 15 years after inclusion
  Beck Depression Inventory (BDI) (total score)
Response to treatment for each therapeutic sequence | every 4-6 months for 15 years after inclusion
  RECIST 1.1 or iRECIST assessment
Response to treatment for each therapeutic sequence | every 4-6 months for 15 years after inclusion
  biological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mario CAMPONE, MD, PhD, Principal Investigator — Institut de Cancerologie de l'Ouest
Locations (2):
- France (2):
  - Institut de Cacerologie de l'ouest - site Paul Papin, Angers
  - Institut de cancerologie de l'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Colombie M, Jezequel P, Rubeaux M, Frenel JS, Bigot F, Seegers V, Campone M. The EPICURE study: a pilot prospective cohort study of heterogeneous and massive data integration in metastatic breast cancer patients. BMC Cancer. 2021 Mar 31;21(1):333. doi: 10.1186/s12885-021-08060-8. PMID 33789635